CLINICAL TRIAL: NCT06101641
Title: Effect of Shellac Nail Polish Application on Pulse Oximetry Measurements in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other); Necmettin Erbakan University (Other); Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Research Assistant, Tarsus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TU-BOZKUL-005
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy Individuals; Shellac Nail Polish; Oxygen Saturation; Nursing; Perioperative Care

STUDY DESIGN:
Intervention Model Description: This study is a prospective, self-controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXPERIMENTAL AND CONTROL GROUP (Other): Participants who meet the inclusion criteria of the study will be informed about the research by the researchers and will be included in the study on a voluntary basis and their written permissions will be obtained. Firstly, the personal information of the participants will be recorded in the data collection form. The middle finger of the left hand of each participant will be the experimental group and the little finger will be the control group. After the shellac nail polish is applied to the middle finger of the left hand, SpO2 and pulse values will be measured by pulse oximetry from the left hand middle finger and little finger of the participant and recorded in the data form. At the end of the study, SpO2 and pulse values before and after the shellac nail polish application will be compared.
  Interventions: Other: Shellac nail polish application

INTERVENTIONS:
Other: Shellac nail polish application — The middle finger of the left hand of each participant will be the experimental group and the little finger will be the control group. After the shellac nail polish is applied to the middle finger of the left hand, SpO2 and pulse values will be measured by pulse oximetry from the left hand middle finger and little finger of the participant
  Other Names: Control group: Non-applied shellac nail

SUMMARY:
The aim of this study was to determine the effect of shellac nail polish application on pulse oximetry measurements in healthy subjects. This study was planned as a prospective, self-controlled clinical research to determine the effect of shellac nail polish application on SpO2 and pulse values in healthy people. The population of the study will consist of women who had shellac nail polish application in a private beauty centre between June 2023 and December 2023. The minimum required sample size was calculated as 162 in G*Power (3.1.9.2) programme (α=0.05 (two-way), 1-β=0.95). The data will be collected with the data collection form prepared in line with the literature. Firstly, the personal information of the participants will be recorded in the data collection form. The middle finger of the left hand of each participant will be the treatment group and the little finger will be the control group. After the shellac nail polish is applied to the middle finger of the left hand, SpO2 and pulse values will be measured simultaneously with a pulse oximeter from the left hand middle finger and little finger of the participant and recorded on the data form. The data obtained from the study will be analysed using SPSS (Statistical Package for Social Sciences) for Windows 26.0 software.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of shellac nail polish application on pulse oximetry measurements in healthy subjects. This study was planned as a prospective, self-controlled clinical research to determine the effect of shellac nail polish application on SpO2 and pulse values in healthy people. The population of the study will consist of women who had shellac nail polish application in a private beauty centre between June 2023 and December 2023. The minimum required sample size was calculated as 162 in G*Power (3.1.9.2) programme (α=0.05 (two-way), 1-β=0.95). The data will be collected with the data collection form prepared in line with the literature. On this form, the age of the individual, the color of the shellac nail, smoking status, and the SpO2 and pulse values measured by pulse oximetry from the little and middle finger will be recorded. SpO2 and pulse rates will be measured with a calibrated Jumper pulse oximeter. Since the shellac nail and non-shellac nail will be measured at the same time, two of the same brand pulse oximeter devices will be provided. Volunteers who meet the inclusion criteria of the research will be informed about the research and will be included in the research on a voluntary basis and their written consent will be obtained. Firstly, the personal information of the participants will be recorded in the data collection form. The middle finger of the left hand of each participant will be the treatment group and the little finger will be the control group. After the shellac nail polish is applied to the middle finger of the left hand, SpO2 and pulse values will be measured simultaneously with a pulse oximeter from the left hand middle finger and little finger of the participant and recorded on the data form. The data obtained from the study will be analysed using SPSS (Statistical Package for Social Sciences) for Windows 26.0 software. Mean and standard deviation will be used in the evaluation of the data. Statistical significance will be accepted as p<0.05 (95% confidence interval).

ELIGIBILITY:
Inclusion Criteria:

* No communication problems,
* With full left-hand fingernails,
* No structural problems such as clubbing,
* Body temperature ≥ 36- <37.5 ºc,
* SpO2 value ≥ 95%,
* Capillary refill ≤ 2 seconds,
* Who volunteered to participate in the research,
* No psychiatric or physical illness that prevents communication,
* Without circulatory problems such as Reynauld syndrome and peripheral arterial disease,
* Without anaemia,
* No respiratory diseases such as chronic obstructive pulmonary disease and asthma
* Becoming a woman

Exclusion Criteria:

* Communication problems,
* Incomplete left fingernails,
* Structural problems like sticky fingers,
* Body temperature ≥ 36- < 37.5 ºc,
* SpO2 value <95%,
* Capillary refill >2 seconds,
* Not volunteering to participate in the research,
* Psychiatric or physical illness that prevents communication,
* With circulatory problems such as Reynauld syndrome and peripheral arterial disease,
* Anaemia
* Respiratory diseases such as chronic obstructive pulmonary disease and asthma
* Not being of the female gender

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
SpO2 value | 6 months
  Data collection form: After the shellac nail polish was applied to the middle finger of the left hand, SpO2 values were measured and recorded by pulse oximetry from the left hand middle finger and little finger of the participant.
Pulse value | 6 months
  Data collection form: After the shellac nail polish was applied to the middle finger of the left hand, pulse values were measured and recorded by pulse oximetry from the left hand middle finger and little finger of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, Assoc. Dr., Principal Investigator — Mersin University; SERPİL YÜKSEL, Assoc.Dr., Principal Investigator — NECMETTİN ERBEKAN UNIVERSITY; AYŞENUR SERBEST BAZ, Principal Investigator — Mustafa Kemal University
Locations (1):
- Tarsus University, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deniz Dogan S, Karacay Yikar S, Arslan S, Nazik E. The Effect of Nail Polish and Henna on the Measures of Pulse Oximeters in Healthy Persons. J Perianesth Nurs. 2021 Oct;36(5):532-535. doi: 10.1016/j.jopan.2020.10.013. Epub 2021 Apr 26. PMID 33926803
- [Background] Ballesteros-Pena S, Fernandez-Aedo I, Picon A, Lorrio-Palomino S. [Influence of nail polish on pulse oximeter readings of oxygen saturation: a systematic review]. Emergencias. 2015 Oct;27(5):325-331. Spanish. PMID 29087059
- [Background] An R, An R. Comparative Study of Spo2 in all the Fingers of the Hands Measured by Pulse Oximeter. J Assoc Physicians India. 2022 Apr;70(4):11-12. PMID 35443453
- [Background] Hakverdioglu Yont G, Akin Korhan E, Dizer B. The effect of nail polish on pulse oximetry readings. Intensive Crit Care Nurs. 2014 Apr;30(2):111-5. doi: 10.1016/j.iccn.2013.08.003. Epub 2013 Sep 17. PMID 24054173
- [Background] Yeganehkhah M, Dadkhahtehrani T, Bagheri A, Kachoie A. Effect of Glittered Nail Polish on Pulse Oximetry Measurements in Healthy Subjects. Iran J Nurs Midwifery Res. 2019 Jan-Feb;24(1):25-29. doi: 10.4103/ijnmr.IJNMR_176_17. PMID 30622574